CLINICAL TRIAL: NCT06214988
Title: SELective Defunctioning Stoma Approach in Low Anterior Resection for Rectal Cancer (SELSA): a Prospective Study With a Nested Randomised Clinical Trial
Brief Title: Selective Defunctioning Stoma in Low Anterior Resection for Rectal Cancer
Acronym: SELSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Umeå University (Other); Lund University (Other); Göteborg University (Other); Ersta Hospital, Sweden (Other); Copenhagen University Hospital at Herlev (Other); Linkoeping University (Other Government); Oslo University Hospital (Other); Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Pamela Buchwald, associate professor, senior consultant surgeon, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0437-01
Record Dates: First submitted 2023-12-17; First posted 2024-01-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Rectal Cancer
Keywords: anterior resection; defunctioning stoma; selective approach
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Observational trial with nested randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- selective approach to defunctioning stoma (Experimental): With randomisation to this experimental arm (selective approach), no defunctioning stoma is constructed.
  Interventions: Procedure: selective approach defunctioning stoma
- routine use of defunctioning stoma (No Intervention): With randomisation to this control arm (systematic approach), a defunctioning stoma is constructed using the marked stoma site. A loop ileostomy is fashioned using an ileal loop close to the ileocecal valve, while a loop colostomy can be derived from either the transverse or a redundant left colon.

INTERVENTIONS:
Procedure: selective approach defunctioning stoma — With randomisation to this experimental arm (selective approach), no defunctioning stoma is constructed.
  Arms: selective approach to defunctioning stoma

SUMMARY:
The goal of this observational trial with a nested randomized controlled trial is to investigate a selective approach of defunctioning stoma in low anterior resection in rectal cancer patients. The primary outcome is a hybrid so-called textbook outcome; stoma-free survival at two years without major LARS, reflecting a functionally appropriate outcome after low anterior resection for rectal cancer. Secondary outcomes include anastomotic leakage, postoperative mortality, reinterventions, stoma-related complications, quality of life measures, LARS, and permanent stoma rate up to two years after index surgery.

DETAILED DESCRIPTION:
Systematic use of defunctioning stoma after low anterior resection for rectal cancer has been shown to reduce symptomatic anastomotic leakage and associated interventions. However, accumulating data suggest that this comes at the price of worse bowel dysfunction, a higher rate of permanent stomas and kidney injury. We aim to study whether a selective strategy of defunctioning stoma use might lead to fewer adverse consequences, while still being safe for patients.

This is a multicentre international prospective trial including a non-blinded randomised clinical trial. All patients with a primary rectal cancer planned for low anterior resection with colorectal or coloanal anastomosis are eligible. Patients enter a prospective observational study, in which a randomised clinical trial is nested. Patients eligible for randomisation are aged below 80 years, have an American Society of Anesthesiologists' fitness grade I or II, have no unresected distant disease, and have a predicted lower risk of anastomotic leakage. Patients will be randomised 1:1 to either an experimental arm with no defunctioning stoma or to a control arm with a defunctioning stoma. The randomisation is computer-generated with a concealed sequence and stratified by participating hospital and radiotherapy use. The main outcome is the composite measure of 2-year stoma-free survival without major low anterior resection syndrome (LARS). Secondary outcomes include anastomotic leakage, postoperative mortality, reinterventions, stoma-related complications, quality of life measures, LARS, and permanent stoma rate up to two years after index surgery. To be able to state superiority of any study arm regarding the main outcome, with 90% statistical power and assuming 25% attrition, we aim to enrol 212 patients.

This study has been approved by Ethical Review Authority in Sweden (2023-04347-01) and seeks permission in Norway and Danmark, respectively. The results will be disseminated through patient associations, popular science, the broader medical community, and conventional scientific channels.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with rectal cancer planned for a low anterior resection with anastomosis by TME with any surgical approach

Additional inclusion criteria for randomised part of the study:

* Patients aged less than 80 years
* Patients with American Society of Anesthetists' (ASA) fitness grade I or II as determined by the anaesthesiologist or the surgeon
* Patients without clear radiological signs of distant disease before rectal cancer surgery (previous metastatic surgery is no exclusion criterion)
* Anastomotic leak risk score of 0-1
* Willingness to be randomised

Exclusion Criteria:

* Insufficient command of Swedish, Norwegian, Danish or English to understand questionnaires or consent
* Emergency rectal resection (tumour resection due to large bowel obstruction, perforation, etc)
* Pregnancy or breastfeeding Additional exclusion criteria for randomised part of the study
* Previous pelvic irradiation (due to e.g. gynaecological or urological cancer)
* Preoperative tumour perforation or pelvic sepsis
* Beyond TME surgery and/or concurrent resection of other organ
* Concurrent corticosteroid treatment (prednisone-equivalent dosage ≥10 mg daily)
* Planned postoperative chemotherapy
* Smoking not completely ceased four weeks before surgery
* Excessive alcohol consumption with social and medical consequences (as judged by the surgeon in charge) Intraoperative exclusion criteria for randomised part of the study

  ->2 staple firings for rectal transection
* Intraoperative blood loss ≥250 ml for minimally invasive surgery
* Intraoperative blood loss ≥500 ml for open or converted surgery
* More than one intraabdominal anastomosis performed
* Incomplete doughnuts
* Air-leak test positive
* Any significant intraoperative adverse event at the discretion of the operating surgeon (e.g. ureterotomy, bowel or tumour perforation, major medical event - pulmonary embolism, cardiac arrhythmia) (Gawria, 2022)
* TME with anastomosis ultimately not done

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
textbook outcome; stoma-free survival at two years without major LARS | 2 year
  extant stoma, alive, and a LARS score at 30 or lesn has stabilised as well for those without a stoma in situ.
  no extant stoma, alive, and a LARS score at 30 or less at the time point two years after the anterior resection.

SECONDARY OUTCOMES:
Anastomotic leakage | 1,3,12 and 24 months
  ISREC grading
Complications | 1,3,12 and 24 months
  Clavien-Dinco
Length of hospital stay | until discharge within 90 days
  total days in hospital
Postoperative mortality | 3 months
  death
Major Low Anterior Resection Syndrome | 12 and 24 months
  domain score scale 0-42 points, >30 points indicate a bad functional outcome i.e. major LARS
Quality of life by European Organization for Research and Treatment of Cancer- ColoRectal 29 (EORTC-CR29) | 12 and 24 months
  EORTC-CR29 domain scores in scales 0-100 points, a high score for the global health status /quality of life represents a high quality of life, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Quality of Recovery-15 Swedish (QoR15swe) | 1 month
  Difference from baseline in total score 0-150 points, higher value indicating faster recovery
Adjuvant chemotherapy for high-risk patients | 12 months
  Clinical assessment categorisation
Renal function | 12 and 24 months
  Creatinine (mg/L)
Stay out of hospital | 24 months
  total days of alive and out of hospital
Stoma in situ | 24 months
  proportion
Recurrence (local and distant) | 36 and 60 months
  Clinical assessment categorisation
Overall survival | 36 and 60 months
  Clinical assessment categorisation
Quality of life by European Organization for Research and Treatment of Cancer- Cancer30 (EORTC-C30) | 12 and 24 months
  EORTC-C30 domain scores in scales 0-100 points, a high score for the global health status /quality of life represents a high quality of life, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Buchwald, MD PhD, Principal Investigator — Skåne University Hospital, Lund University; Martin Rutegård, MD PhD, Principal Investigator — Umeå University Hospital, Umeå University Hospital
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Unidentified raw data may be shared upon request.
Supporting Information: Study Protocol, SAP
Time Frame: When study complete including primary and secondary endpoints.

REFERENCES:
- [Derived] Rutegard M, Lindskold M, Jorgren F, Landerholm K, Matthiessen P, Forsmo HM, Park J, Rosenberg J, Schultz J, Seeberg LT, Segelman J, Buchwald P. SELective defunctioning Stoma Approach in low anterior resection for rectal cancer (SELSA): Protocol for a prospective study with a nested randomized clinical trial investigating stoma-free survival without major LARS following total mesorectal excision. Colorectal Dis. 2025 Feb;27(2):e70009. doi: 10.1111/codi.70009. PMID 39887540

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT06214988/Prot_SAP_000.pdf